CLINICAL TRIAL: NCT04841057
Title: Biometabolic Outcomes After Weight Loss Surgery: An Individualized Approach
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Andrew Wheeler, Assistant Professor of Surgery, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2032062
Record Dates: First submitted 2021-04-08; First posted 2021-04-12 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Obesity, Morbid; Metabolic Syndrome; NASH - Nonalcoholic Steatohepatitis
Keywords: gastric bypass; intestinal bypass; gut microbiome; microRNA; enteroendocrine hormones; weight recidivism; biliopancreatic limb
MeSH Terms: conditions — Obesity, Morbid; Metabolic Syndrome; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: Patients undergoing gastric bypass
Who Masked: Participant
Masking Description: Blinded to participant at time of surgery. Randomization during operation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard BP limb length (Experimental): 50 cm BP limb length
  Interventions: Procedure: 50 cm BP limb length
- Medium BP limb length (Experimental): 100 cm BP limb length
  Interventions: Procedure: 100 cm BP limb length
- Long BP limb length (Experimental): 150 cm BP limb length
  Interventions: Procedure: 150 cm BP limb length

INTERVENTIONS:
Procedure: 50 cm BP limb length — 50 cm biliopancreatic limb length
  Arms: Standard BP limb length
Procedure: 100 cm BP limb length — 100 cm biliopancreatic limb length
  Arms: Medium BP limb length
Procedure: 150 cm BP limb length — 150 cm BP limb length
  Arms: Long BP limb length

SUMMARY:
Variable outcomes after weight loss surgery are likely attributable to complex, poorly understood mechanisms. Due to the significant impact that morbid obesity has on a patient's health, successful management of obesity and its related comorbid medical conditions is important and thus necessitates continued improved therapies for treating obesity. Although the mechanisms of weight loss after surgical intervention are poorly understood, improved understanding of molecular and metabolic changes that occur after weight loss surgery may offer the ability to provide targeted precision therapy for patients with morbid obesity undergoing surgical therapy. In this proposal, the investigators will combine a clinical trial whereby modifications to the gold-standard for weight loss surgery, the gastric bypass, are evaluated while simultaneously measuring molecular and metabolic changes that occur in response to these weight loss procedures. Through creating variable lengths of bypass intestine after gastric bypass, the investigators will be able to determine the effect of malabsorption on clinical outcomes and mechanisms involved in weight loss after gastric bypass. The investigators will also use two control groups. One will be a surgical weight loss control group and consist of patients undergoing a laparoscopic sleeve gastrectomy, a non-intestinal bypass procedure. The other group will consist of patients having non-surgical weight loss therapy. To asses metabolic changes that occur in response to surgical weight therapy and specifically intestinal bypass and malabsorption, the investigators will examine changes in the gut microbiome and plasma gut enteroendocrine hormones. To evaluate molecular pathways that are impacted as a result of gastric bypass and malabsorption, the investigators will measure circulating microRNAs (miRNAs) in the blood. Measurement of miRNAs will provide data on an easily measurable molecular marker for each treatment group. This is a first step in translational exploration of mechanisms of weight loss after surgery by evaluating both clinical and molecular/metabolic outcomes and begin an explorative process towards creating an individualized approach to improving outcomes after weight loss surgery.

DETAILED DESCRIPTION:
Outcomes after weight loss surgery are quite variable with some patients regaining a significant amount of weight in the postoperative period. Increasing evidence suggests gastric bypass leads to weight loss and improvement in associated metabolic illness through mechanisms other than just restriction and malabsorption and may include circulating bile acids, gut hormones, genetic/epigenetic variability, changes in gut microbiota as well as other mechanisms. Whether modifications to bypassed intestine length may improve outcomes after gastric bypass has not been adequately studied with inconsistent results in the literature. Whether increasing the amount of bypassed intestine may positively amplify the multi-factorial mechanisms involved in successful weight loss has not been studied.

The primary goal of the research is to determine if increasing the amount of bypassed intestine during gastric bypass surgery improves outcomes and effects molecular and metabolic changes that may impact outcomes after gastric bypass. The proposed research will evaluate not only biologic mechanisms of weight loss and correlation between these mechanisms and successful weight loss but also investigate the role intestinal bypass has on molecular and metabolic mechanisms involved in effective weight loss therapy. Regardless if weight loss outcomes are similar in patients with different lengths of bypassed intestine, the role of the gut in gastric bypass will be investigated through evaluation of gut microbiota, circulating miRNAs and gut hormones, three mechanisms thought to play a role in the effectiveness of the gastric bypass for weight loss surgery.

Aim 1: Determine if increasing length of bypassed intestine leads to improved clinical outcomes after gastric bypass. A randomized-controlled trial design will be used with patients randomized to variable lengths of bypassed intestine when undergoing gastric bypass. A randomized trial will help avoid procedure selection bias. Surgical and non-surgical control groups will consist of patients having sleeve gastrectomy (non-intestinal bypass surgical control) and those undergoing best non-surgical, medical therapy. Primary outcomes measured will include weight loss and relief of medical comorbidities of obesity specifically diabetes and dyslipidemia. Secondary outcomes include complications related to malabsorption.

Aim 2: Measure gut hormone changes after increased intestinal bypass during gastric bypass. The investigators will measure gut hormones after variable amounts of intestinal bypass to determine the role of intestinal bypass in improvement of gut hormone production that affects metabolism, hunger and possibly weight loss. Blood collected from patient's in Aim 1 will be used to measure gut hormone levels which will then be correlated to clinical outcomes.

Aim 3: miRNA profiling in patients having gastric bypass with variable intestinal bypass lengths. The investigators will perform miRNA arrays on plasma from patients from Aim 1 to determine possible pathways impacted by weight loss and in particular increased intestinal bypass lengths in patients undergoing gastric bypass. The variable expression of miRNA will also be correlated to weight loss outcomes and metabolic disease improvement in the surgical patients.

Aim 4: Measure variation in gut microbiome due to increased intestinal bypass during gastric bypass. The investigators will examine the impact of weight loss and variable intestinal bypass lengths during gastric bypass on the gut microbiome. This will be determined through collection of stool samples preoperatively as well as postoperatively in patients having weight loss surgery. Samples will be collected from patients in Aim 1 above. Sleeve gastrectomy patients will be used to determine the impact of surgical weight loss on gut microbiome and variation in intestinal bypass lengths will provide insight into the role of bypassed intestine in the effects of gastric bypass on changes in gut microbiota after weight loss surgery. Through correlation with clinical outcomes the investigators will be able to determine any association with weight loss and relief of metabolic disease when the gut microbiota are modified after weight loss surgery.

Approach

Protocol Aim 1: Determine if increasing length of bypassed intestine leads to improved clinical outcomes after gastric bypass.

Primary outcomes will include weight loss and relief of medical comorbidities of obesity, in particular diabetes and dyslipidemia. Secondary outcomes include determining complications that occur such as protein calorie malnutrition, vitamin and micronutrient deficiencies and chronic diarrhea.

1a. Randomization of patients and surgical technique. A total of five groups will be used. The surgical control group will consist of patients having a laparoscopic sleeve gastrectomy as described below under procedure descriptions. The non-surgical control group will include patients undergoing best medical therapy through our medical weight loss program. The other three groups will be randomized through a sealed-envelope method. The assigned group will be in a sealed envelope and the patient will be blinded to the treatment group that they are assigned to. Patients will be randomized to variable lengths of intestinal bypass during performance of a laparoscopic Roux-en-Y gastric bypass. See description of procedure below. These groups will function to examine the impact of increasing lengths of bypassed small intestine through modifications of the BPL length. The following three groups will be utilized:

1. Alimentary limb length 100 cm and biliopancreatic limb length (true bypassed intestinal length) of 50 cm
2. Alimentary limb length 100 cm and biliopancreatic limb length (true bypassed intestinal length) of 100 cm
3. Alimentary limb length 100 cm and biliopancreatic limb length (true bypassed intestinal length) of 150 cm Sample size for randomization to the three gastric bypass groups will be approximately 75 patients in each group. 75 sleeve gastrectomy patients will also be included. Sample size was determined based on previously published literature. The total number of these patients will be used only for the clinical portion of the study. Sample size for this pilot study for each of the gut hormone assays, gut microbiome analyses and miRNA arrays will be 15 subjects in each group. This will include 15 patients selected from each of the groups of randomized gastric bypass patients, the sleeve gastrectomy group, and the medical control group for a total of 75 patients. Each patient will have stool and blood collected at pre-treatment (surgical or non-surgical therapy), 6 months post therapy and 12 months post therapy.

Surgical Procedure A gastric bypass will be performed using our standard technique. In brief, all procedures will be performed laparoscopically as is standard practice. Specifically at our institution, the gastric pouch will be constructed with a linear stapler approximately 5 cm long and 3 cm wide. The gastrojejunostomy anastomosis will be constructed either with a 25 mm circular stapler or a linear stapler. The linear stapler common gastroenterotomy will be closed in a running 2 layer manner to narrow to approximately 13-15 mm. The jejunojejunostomy will be created with a liner stapler after creation of BPL length of 50 cm, 100 cm or 150 cm and an alimentary limb length of 100 cm which will be connected to the gastric pouch via the gastrojejunostomy. The remaining small bowel, which will represent the common small bowel channel will also be measured. Measurements will be achieved using premeasured markings on a laparoscopic grasper used to handle the small intestine.

Patients undergoing a sleeve gastrectomy will serve as the control group in order to determine the effect that intestinal bypass has on the measured outcomes. The sleeve gastrectomy is performed laparoscopically to resect and remove approximately 80% by volume of the outer portion of the stomach. At our institution, specifically the sleeve gastrectomy is performed using multiple firings of a laparoscopic stapler using a bougie as an intraluminal template for sizing purposes. The bougie is either 36 or 40 French per our usual practice.

2a. Sample collection preoperatively and postoperatively for metabolic and molecular studies.

Sample Collection

Samples will be collected and processed by the OneHealth Biorepository or other on site research laboratory. The following samples will be collected in each patient:

1. Blood: will be collected at a preoperative time point then at 6 months and 12 months postoperatively. The blood will be drawn by MU Health Care laboratories or associated research personnel and transported by courier per standard protocol to the OneHealth Biorepository or other research lab. It will be fractionated into its components and plasma collected and stored at -80℃ as previously described.
2. Stool: Stool samples will be collected by patients at home using provided kits and mailed to the OneHealth Biorepository or other affiliated research lab and stored, as previously described. Samples will be aliquoted and stored at -20℃.

3a. Prospective collection of clinical data. Weight related data will be collected to determine effectiveness of weight loss operations. Weight data collected will include high weight when entering the weight loss surgery program, immediate preoperative weight collected on day of operation and postoperative weights at 1 week, 1 month, 3 months, 6 months and 12 month follow-up appointments. Additional outcomes collected will include presence of diabetes mellitus with glycated hemoglobin (HgbA1C) levels measured preoperatively and at 6 and 12 months postoperatively Remission of diabetes will be considered if the patient is off all anti-diabetic medications with a normal HgbA1C. Presence of preoperative dyslipidemia will also be documented to include abnormalities of LDL cholesterol, HDL cholesterol and triglyceride levels. Remission of dyslipidemia will be considered if preoperative abnormal levels of LDL and HDL cholesterol and triglycerides return to normal in the absence of lipid-lowering agents.

Aim 2: Measure gut hormone changes after increased intestinal bypass during gastric bypass Millipore Human Metabolic Hormone Magnetic Bead Panel - Metabolism Multiplex Assay will be used to investigate a panel of gut hormones including GLP-1, GIP, leptin, PYY, and ghrelin. Plasma from 15 patients from each group (as described above) for a total of 75 total patients will be examined. Hormone levels in the plasma will be measured. Data will be analyzed both for intergroup differences as well as correlation with clinical outcomes will be performed.

Aim 3: miRNA profiling in patients having gastric bypass with variable intestinal bypass lengths 15 patients from each group (as described above) for a total of 75 total patients will be examined. Plasma will be used to perform Affymetrix miRNA arrays to measure expression of all currently known miRNA. Corresponding pathways that miRNA affect will be identified using publicly available databases. Differences in miRNA expression between treatment groups will be compared. Differential levels of expression of miRNA will also be compared to clinical outcomes.

Aim 4: Measure variation in gut microbiome due to increased intestinal bypass during gastric bypass.

Stool samples will be collected as described above. They will be stored in the OneHealth Biorepository or other laboratory until processing. 15 patients from each group (as described above) for a total of 75 total patients will be examined. Composition of microbiota in each group will be determined as previously described. Comparison between treatment groups will be performed. Correlation to clinical outcome variables will be determined

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18
2. Body mass index of 40-60 kg/m2
3. Meet insurance criteria, as set forth by the patient's insurance policy, to qualify for coverage for weight loss surgery
4. Planned laparoscopic Roux-en-Y gastric bypass
5. Willingness to have blood collected before and after surgical procedure at defined points and collect and mail stool sample before operation and at defined post-operative time points.

Exclusion Criteria:

1. Age less than 18
2. Patient fails to fulfill insurance mandated criteria
3. Unwilling to be randomized to variable length to gastric bypass or unwilling to have blood collected or personally collect and mail in stool sample
4. Unwilling to follow-up at required postoperative visits

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2031-03-01 (Estimated); Study Completion 2031-03-01 (Estimated)

PRIMARY OUTCOMES:
Weight loss after Variable Biliopancreatic Limb Length Bypass | 7 years
  Evaluation of weight loss after modifications to the length of BP limb length
Complications after Variable Biliopancreatic Limb Length Bypass | 7 years
  Evaluation of weight loss after modifications to the length of BP limb length

SECONDARY OUTCOMES:
MicroRNA expression after Variable Biliopancreatic Limb Length Bypass | 7 years
  measurement of circulating microRNA expression in treatment groups
Gut microbiome changes after Variable Biliopancreatic Limb Length Bypass | 7 years
  measurement of circulating microRNA expression in treatment groups
Gut enteroendocrine changes after Variable Biliopancreatic Limb Length Bypass | 7 years
  measurement of circulating microRNA expression in treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Wheeler, MD, Principal Investigator — University of Missouri-Columbia, Department of Surgery
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Only deidentified samples and clinical data with all HIPAA identifiers will be shared with any other researchers
Supporting Information: Study Protocol, SAP
Time Frame: Data will only be made available on a case by case data and provided in a deidentified manner
Access Criteria: Data must be deidentified and data must be requested from the PI listed